CLINICAL TRIAL: NCT02229747
Title: Randomized, Open-label, Controlled Trial to Assess the Clinical Efficacy and Safety of Meloxicam Suspension 0.25 mg/kg/Day Once a Day, Versus Diclofenac 1 mg/kg/Day Twice a Day or Nimesulide 4 mg/kg/Day Twice a Day, for Five Days in the Treatment of Patients With Acute, Non-bacterial Pharyngitis, Pharyngotonsillitis or Laryngitis
Brief Title: Efficacy and Safety of Meloxicam Suspension Versus Diclofenac Suspension or Nimesulide Suspension in Patients With a Diagnosis of Acute, Non-bacterial Pharyngitis, Pharyngotonsillitis or Laryngitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107.250
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-07

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Meloxicam; Diclofenac; nimesulide

ARMS (3):
- Meloxicam suspension (Experimental)
  Interventions: Drug: Meloxicam
- Diclofenac suspension (Active Comparator)
  Interventions: Drug: Diclofenac
- Nimesulide suspension (Active Comparator)
  Interventions: Drug: Nimesulide

INTERVENTIONS:
Drug: Meloxicam
  Arms: Meloxicam suspension
Drug: Diclofenac
  Arms: Diclofenac suspension
Drug: Nimesulide
  Arms: Nimesulide suspension

SUMMARY:
The objective of this study was to assess the clinical efficacy and safety of meloxicam suspension 0.25 mg/kg/day once a day, versus diclofenac suspension 1 mg/kg/day twice a day or nimesulide suspension 4 mg/kg/day twice a day, after five days of treatment in patients with a diagnosis of acute, non-bacterial pharyngitis, pharyngotonsillitis or laryngitis

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders between 2 and 8 years old
* Outpatients, with onset of symptoms not more than 72 hours prior to presentation, patients with acute non-bacterial pharyngitis or pharyngotonsillitis diagnosed according to the following criteria:

  * Spontaneous pharyngeal pain, pharyngeal pain upon swallowing, pharyngeal and/or tonsillar hyperemia, absence of purulent plaques, pharyngeal smear negative for ß-hemolytic Streptococcus or Strepto Test® and Treatment with an Non-steroidal anti-inflammatory drugs (NSAID) required or recommended

Exclusion Criteria:

* Known or suspected hypersensitivity to study medications or NSAID's
* Pharyngeal smear positive for ß-hemolytic Streptococcus
* treatment with antimicrobials prior to enrolment in the study
* Chronic infection, infectious mononucleosis, peptic ulcer disease that has been active in the previous 6 months
* Asthma
* nasal polyps
* angioneurotic edema or urticaria after the administration of aspirin or NSAID's
* Concomitant treatment with anticoagulants (including heparin), lithium or methotrexate
* Concomitant administration of other NSAID's (including high dose aspirin) or analgesics, except authorized rescue drugs
* Administration of any NSAID during the three previous days or of analgesics within six hours prior to the administration of the first study drug dose
* Treatment with corticosteroids at the time of enrollment or within the two previous months
* Known liver, renal or hematological disease
* Participation in another clinical trial during the study period or during the previous month
* Previous enrollment in this study
* Inability to comply with the protocol
* Suspected acute bacterial pharyngitis or pharyngotonsillitis (under the following clinical criteria):

  * Clinical presentation characterized by a rapid onset, very high fever (>38.5°C), severe pharyngeal pain, cervical adenopathy, intense headache, purulent pharyngeal plaques, evidence of peritonsillar abscess or phlegmon

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2001-08; Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Change in spontaneous pharyngeal pain | baseline, 5 days
Change in pharyngeal pain on deglutition (dysphagia) | baseline, 5 days
Change in pharyngeal hyperemia | baseline, 5 days
Change in systemic manifestations (fever, adenomegaly and general malaise) | baseline, 5 days
Incidence of adverse events | baseline, 5 days